CLINICAL TRIAL: NCT05647005
Title: The Effect of Classical and Harp Music Practice on Physiological Parameters, Cerebral Oxygenation and Comfort in Premature Infants: A Randomized Controlled Study
Brief Title: The Effect of Classical and Harp Music Practice on Premature Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Selcuk University (Other)
Responsible Party: Principal Investigator, Sevinc Akkoyun, lecturer (Phd), Selcuk University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2022/48
Record Dates: First submitted 2022-12-03; First posted 2022-12-12 (Actual); Last update posted 2024-04-02 (Actual); Status verified 2024-03

CONDITIONS: Music; Premature Infant; Cerebral Oxygenation; Comfort
Keywords: Classical music; Harp Music; Premature infant; Cerebral Oxygenation; Physiological Parameters; Comfort
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Intervention Model Description: It is a parallel, three-group randomized controlled trial with a prospective, pretest, posttest experimental design.
Who Masked: Participant
Masking Description: Single (Participant, outcomes assessor)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Experiment 1: Classical music (Experimental): A total of 15 sessions of music will be applied to this group, two or three days a week, on different days, 3 sessions a day. The sessions will be in the form of listening to classical music for 30 minutes after the babies are fed.
  Interventions: Other: Classical music
- Experiment 2: Harp music (Experimental): A total of 15 sessions of music will be applied to this group, two or three days a week, on different days, 3 sessions a day. Sessions will be in the form of listening to harp music for 30 minutes after the babies are fed.
  Interventions: Other: Harp music
- Control (No Intervention): Premature babies in this group will not be interfered with by the newborn nurses for 30 minutes after feeding without any voice intervention.

INTERVENTIONS:
Other: Classical music — A total of 15 sessions of music will be applied to this group, two or three days a week, on different days, 3 sessions a day. Sessions will be in the form of listening to classical music for 30 minutes after the babies are fed.
  Arms: Experiment 1: Classical music
Other: Harp music — A total of 15 sessions of music will be applied to this group, two or three days a week, on different days, 3 sessions a day. Sessions will be in the form of listening to harp music for 30 minutes after the babies are fed.
  Arms: Experiment 2: Harp music

SUMMARY:
Aim of the study is to determine the effects of classical and harp music practice on physiological parameters (heart rate, respiratory rate and oxygen saturation value), cerebral oxygenation value (rSO2) and comfort of premature infants.

It is a parallel, three-group randomized controlled trial with a prospective, pretest, posttest experimental design. The study will be carried out in Selcuk University Medical Faculty Hospital Neonatal Intensive Care Unit (NICU). A total of 84 premature babies will be included in the study, including the group to be listened to classical music (n=28), the group to be listened to harp music (n=28), and the control group (n=28). Triple blocks were created in the computer environment so that the premature infants to be included in the study could be assigned to three study groups using the balanced block randomization method (randomization.com). The randomization will be hidden from the researcher conducting the trial until the administration begins. The researcher will be given 84 envelopes and will begin to open the envelopes when they meet the baby. The researcher will learn which group each baby is in just before the application. Data collection tools; newborn Descriptive Information Form, physiological parameter and rSO2 follow-up form, and Premature infant comfort scale. The rSO2 value will be measured with the NIRS monitor. During the data collection phase, the purpose of the study will be explained to the parents of the premature infants by the researcher first, and informed about the study and consent will be obtained from the parents who agreed to participate in the study through the "Informed Voluntary Consent Form". To venture groups (classical and harp music); After feeding, a music box and a decibel meter will be placed in the incubator and classical music will be turned on at 50-55 dB. Just before the music is played, the premature infants physiological parameters, rSO2 and comfort level will be evaluated and recorded. For 30 minutes, music will be played to the baby according to the intervention group (classical and harp music). After 30 minutes, the baby's physiological parameters, rSO2 and comfort level will be evaluated and recorded again. Each session will be held in this way, a total of 15 sessions of music will be applied to thepremature infants, and the baby's physiological parameters, rSO2 and comfort level will be evaluated and recorded before and after each session. The control group is; premature infants in this group are those who take the clinical routine without being exposed to any music. After feeding, the baby's physiological parameters, rSO2 and comfort level will be evaluated and recorded. They will not be exposed to any music and sound for 30 minutes and there will be no intervention. At the 30th minute, the premature infants physiological parameters, rSO2 and comfort level will be evaluated and recorded. Evaluation of the data will be done in the computer environment with the SPSS (Statistical Package for Social Sciences) 22.0 package program. Partial eta squared will be calculated for the effect size and the significance level will be accepted as p<0.05.

DETAILED DESCRIPTION:
Aim of the study is to determine the effects of classical and harp music practice on physiological parameters (heart rate, respiratory rate and oxygen saturation value), cerebral oxygenation value (rSO2) and comfort of premature infants.

It is a parallel, three-group randomized controlled trial with a prospective, pretest, posttest experimental design. The study will be carried out in Selcuk University Medical Faculty Hospital Neonatal Intensive Care Unit (NICU). A total of 84 premature babies will be included in the study, including the group to be listened to classical music (n=28), the group to be listened to harp music (n=28), and the control group (n=28). Triple blocks were created in the computer environment so that the premature infants to be included in the study could be assigned to three study groups using the balanced block randomization method (randomization.com). The randomization will be hidden from the researcher conducting the trial until the administration begins. The researcher will be given 84 envelopes and will begin to open the envelopes when they meet the baby. The researcher will learn which group each baby is in just before the application. Data collection tools; newborn Descriptive Information Form, physiological parameter and rSO2 follow-up form, and Premature infant comfort scale. The rSO2 value will be measured with the NIRS monitor. During the data collection phase, the purpose of the study will be explained to the parents of the premature infants by the researcher first, and informed about the study and consent will be obtained from the parents who agreed to participate in the study through the "Informed Voluntary Consent Form". To venture groups (classical and harp music); After feeding, a music box and a decibel meter will be placed in the incubator and classical music will be turned on at 50-55 dB. Just before the music is played, the premature infants physiological parameters, rSO2 and comfort level will be evaluated and recorded. For 30 minutes, music will be played to the baby according to the intervention group (classical and harp music). After 30 minutes, the baby's physiological parameters, rSO2 and comfort level will be evaluated and recorded again. Each session will be held in this way, a total of 15 sessions of music will be applied to thepremature infants, and the baby's physiological parameters, rSO2 and comfort level will be evaluated and recorded before and after each session. The control group is; premature infants in this group are those who take the clinical routine without being exposed to any music. After feeding, the baby's physiological parameters, rSO2 and comfort level will be evaluated and recorded. They will not be exposed to any music and sound for 30 minutes and there will be no intervention. At the 30th minute, the premature infants physiological parameters, rSO2 and comfort level will be evaluated and recorded. Evaluation of the data will be done in the computer environment with the SPSS (Statistical Package for Social Sciences) 22.0 package program. Partial eta squared will be calculated for the effect size and the significance level will be accepted as p<0.05.

ELIGIBILITY:
Inclusion Criteria:

* Premature babies born between 30-36+6
* Postnatal babies at least 5 days old
* Babies with an APGAR score of 7 and above
* Babies with spontaneous breathing and stable hemodynamics
* No history of surgery

Exclusion Criteria:

* Babies with congenital hearing loss
* Babies using sedatives or muscle relaxants
* Absence of congenital anomalies, metabolic diseases, heart diseases and/or other serious diseases

Ages: 30 Weeks to 37 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 84 (Actual)
Dates: Start 2022-12-01 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
rSO2 level | before the intervention and the end of the intervention (30. minutes)
  rSO2 level change
comfort | before the intervention and the end of the intervention (30. minutes)
  comfort level change

SECONDARY OUTCOMES:
Heart rate | before the intervention and the end of the intervention (30. minutes)
  Heart rate change
Respiration rate | before the intervention and the end of the intervention (30. minutes)
  Respiration rate change
SpO2 level | before the intervention and the end of the intervention (30. minutes)
  SpO2 level change

CONTACTS AND LOCATIONS:
Overall Officials: Fatma Tas Arslan, professor, Study Director — Selcuk University; Tuğba Genç, nurse, Study Chair — Selcuk University
Locations (1):
- Selcuk University, Konya, Selcuklu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
The Effect of Classical and Harp Music Practice on Premature Infants
Supporting Information: Study Protocol
Time Frame: December 2022-July 2023 (7 months)